CLINICAL TRIAL: NCT05320640
Title: A PhaseⅠ/Ⅱ Trial of Chidamide，Decitabine and Immune Checkpoint Inhibitors in Relapsed/Refractory Non-Hodgkin Lymphoma and Advanced Solid Tumors
Brief Title: Study of Chidamide, Decitabine and Immune Checkpoint Inhibitors in R/R NHL and Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-069
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Relapsed/Refractory Non-Hodgkin Lymphoma; Advanced Solid Tumors
Keywords: Relapsed/Refractory Non-Hodgkin Lymphoma; Advanced Solid Tumors; Chidamide; Decitabine; Immune Checkpoint Inhibitors; Chemotherapy free regimen
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Drug: Chidamide10mg/day, day1-4; 20mg/day, day8, 11, 15, 18. Drug: Decitabine10mg/day, day1-5. Drug: Immune Checkpoint Inhibitors（anti-PD1/PD-L1/CTLA4 antibodies）. Physicians will decide which ICIs will be used during treatment.
  Every 3 weeks.
  Interventions: Drug: Chidamide; Drug: Decitabine; Drug: Immune checkpoint inhibitors（anti-PD1/PD-L1/CTLA4 antibodies）

INTERVENTIONS:
Drug: Chidamide — Chidamide is a novel and orally active benzamide class of HDAC inhibitor that selectively inhibits activity of HDAC1, 2, 3 and 10, which can induce tumor-cell apoptosis, suppress cell proliferation and enhance immune surveillance.
Drug: Decitabine — Low-dose decitabine inhibits the activity of DNA methyltransferase, which can increase tumor antigens and HLA expression, enhance antigen processing, promote T cell infiltration, and boost effector T cell function.
Drug: Immune checkpoint inhibitors（anti-PD1/PD-L1/CTLA4 antibodies） — Immune checkpoint inhibitors (ICIs) have emerged as effective therapies for many cancers by promoting the reactivation and restoring function of T cells.

SUMMARY:
This phase I/II trial aims to evaluate safety and efficacy of Chidamide, Decitabine and Immune checkpoint inhibitors in relapsed/refractory Non-Hodgkin Lymphoma and advanced solid tumors.

DETAILED DESCRIPTION:
Chidamide is a novel and orally active benzamide class of HDAC inhibitor that selectively inhibits activity of HDAC1, 2, 3 and 10, which can induce tumor-cell apoptosis, suppress cell proliferation and enhance immune surveillance. Low-dose decitabine inhibits the activity of DNA methyltransferase, which can increase the expression of tumor antigens and HLA molecules, enhance antigen processing, promote T cell infiltration, and boost effector T cell function. Immune checkpoint inhibitors (ICIs) have emerged as effective therapies for many cancers by promoting the reactivation and restoring function of T cells. In conclusion, we speculate that the chemotherapy free regimen of Chidamide, Decitabine and Immune checkpoint inhibitors may explore a new avenue for therapeutic intervention in relapsed/refractory Non-Hodgkin Lymphoma and advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. 16 to 80 years of age.
2. ECOG performance of less than 3.
3. Life expectancy of at least 3 months.
4. Histopathological confirmed Non-Hodgkin Lymphoma and solid tumors.
5. Patients are relapsed/refractory Non-Hodgkin Lymphoma with ineligible for autologous hematopoietic stem cell transplantation.
6. The guidelines（ASCO/CSCO）recommend patients to participate in clinical trials.
7. Subjects must have at least one measureable target lesion.
8. Willingness to provide written informed consent for the study.

Exclusion Criteria:

1. Active, known or suspected autoimmune diseases.
2. Subjects are being treated with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
3. History of severe hypersensitive reactions to other monoclonal antibodies.
4. History of allergy or intolerance to study drug components.
5. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
6. History or concurrent condition of interstitial lung disease of any grade or severely impaired pulmonary function.
7. Uncontrolled intercurrent illness, including ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia) or psychiatric illness/social situations and any other illness that would limit compliance with study requirements and jeopardize the safety of the patient.
8. History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
9. Pregnant or breast-feeding. Women of childbearing potential must have a pregnancy test performed within 7 days before the enrollment, and a negative result must be documented.
10. Vaccination within 30 days of study enrollment.
11. Active bleeding or known hemorrhagic tendency.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 years
  The percentage of patients with CR or PR was determined according to the revised lymphoma efficacy evaluation criteria (Lugano 2014 criteria) and Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Adverse events | 3 years
  Incidence, nature, and severity of adverse events are graded according to the National Cancer Institute Common Terminology Criteria for adverse events (version5.0).

SECONDARY OUTCOMES:
Duration of response (DOR) | 3 years
  Time from the first recording of CR or PR evidence to disease progression or death from any cause was determined according to the revised lymphoma efficacy evaluation criteria (Lugano 2014 criteria) and Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Progression-free survival (PFS) | 3 years
  Time from the date of first administration of the study drug to disease progression or death from any cause.

OTHER OUTCOMES:
Biomarkers predictive of response | 3 years
  Biomarkers from tumor cells, lymphocytes and tumor microenvironment will be assessed for their potential in predicting clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Prfessor, Principal Investigator — Biotherapeutic Department, Chinese PLA General Hospital
Locations (1):
- Biotherapeutic Department, Chinese PLA General Hospital, Beijing, Beijing Municipality, China